CLINICAL TRIAL: NCT06613932
Title: Clinical and Radiographic Assessment of L-PRF, Nanohydroxyapatite Material Combined With L-PRF Scaffold in Vital Pulp Therapy. Treatments in Mandibular First Molars With Closed Apices "Randomized Controlled Trial"
Brief Title: Assessment of L-PRF, Nanohydroxyapatite Combined With L-PRF Using Pulpotomy in Mature Mandibular First Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Nada Ayman El-Sayed Ibraim, principal investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (37)11-2023
Record Dates: First submitted 2024-08-16; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hydroxyapatite (Experimental): using hydroxyapatite as a pulpotomy agent and reviewing its clinical and radiographic performance compared to the other groups
  Interventions: Procedure: pulpotomy
- L-PRF (Experimental): using L-PRF as a pulpotomy agent and assessing the clinical and radiographic result compared to other groups
  Interventions: Procedure: pulpotomy
- L-PRF combined with Nano-hydroxyapatite (Experimental): using the combined material (nanohydroxyapatite mixed to L-PRF ) and assessing the clinical and radiographic result compared to other groups
  Interventions: Procedure: pulpotomy

INTERVENTIONS:
Procedure: pulpotomy — removal of the coronal pulp tissue and preservation of the radicular portion to ensure continuation of growth and vitality of tooth structure
  Other Names: vital pulp therapy

SUMMARY:
Clinical and Radiographic Assessment of L-PRF, Nanohydroxyapatite material combined with L-PRF scaffold in Vital pulp Therapy. Treatments in Mandibular First Molars with Closed Apices, Randomized Controlled Trial.

DETAILED DESCRIPTION:
pulpotomy by using 3 materials. The first group(control group ) uses hydroxyapatite material as a pulpotomy agent, and the second group uses L-PRF as a pulpotomy agent. the third group uses combined material (L-PRF = Nano hydroxyapatite )as a pulpotomy agent .. then assesses the clinical and radiographic result of the 2 interventions group with control group

ELIGIBILITY:
Inclusion criteria:

Patients should be free from any systemic disease. Patients of either gender aged from 15-30. Patients will agree to the consent and will commit to a follow-up period. Soft tissues around the tooth are normal with no swelling or sinus tract. The tooth is restorable tooth has signs and symptoms of irreversible pulpitis of the mature root The tooth doesn't contain any internal or external resorption or periapical lesions.

The tooth should give a positive response to the cold test.

Exclusion criteria:

Pregnant and lactating females. Patients with Mental disturbance. Patients who could/would not participate in a 6-month follow-up. A tooth with immature roots. Patients with necrotic pulp.• tooth with periapical lesions or infections. Soft tissue having fistula or swelling Homoeostasis after 10 minutes can not be controlled after total pulpotomy

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
post operative Pain assessment | 6, 12, 24, 72hours and 7 days after treatment
  Pain evaluations were conducted preoperatively with numerical rating scale ( a verbal or writing determination of a pain level on a scale from 0 to 10, in which 0 represents no pain and 10 represents excruciating pain .

SECONDARY OUTCOMES:
Dentine bridge formation | 12 months post operative
  evaluating the thickness of dentine bridge formed after the procedure by comparing immediate post operative CBCT with the one year follow up scans

CONTACTS AND LOCATIONS:
Overall Officials: wael K hussein, professor, Study Director — future
Locations (1):
- future university in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No